CLINICAL TRIAL: NCT00346684
Title: Rituximab in Primary LPHD (RIPL) - First Line Therapy for Patients With Lymphocyte Predominant Hodgkin´s Disease (LPHD) in Clinical Stage IA Using the Monoclonal Anti-CD20 Antibody Rituximab.
Brief Title: Rituximab in Primary Lymphocyte Predominant Hodgkin´s Disease(RIPL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIPL
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Lymphocyte Predominant Hodgkin´s Lymphoma (LPHD)
Keywords: Lymphoma; LPHD; Rituximab
MeSH Terms: conditions — Lymphoma | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
First line therapy for patients with Lymphocyte predominant Hodgkin´s Disease (LPHD) in clinical stage IA using the monoclonal anti-CD20 antibody rituximab

ELIGIBILITY:
Inclusion Criteria:

* lymphocyte predominant Hodgkin´s lymphoma (histologically proven)
* clinical stage IA (without risk factors: large mediastinal mass, extranodal involvement, ESR > 50mm/h)
* age 18 - 75
* WHO performance status 0-3
* normal organ function
* written informed consent

Exclusion Criteria:

* classical Hodgkin´s lymphoma
* composite lymphoma
* leucocytes < 3000/µl
* thrombocytes < 100.000/µl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-07; Primary Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Principal Investigator — Universitiy of Cologne
Locations (1):
- University of Cologne, Cologne, Germany

REFERENCES:
- [Derived] Eichenauer DA, Plutschow A, Fuchs M, Hartmann S, Hansmann ML, Boll B, von Tresckow B, Borchmann P, Engert A. Rituximab in newly diagnosed stage IA nodular lymphocyte-predominant Hodgkin lymphoma: long-term follow-up of a phase 2 study from the German Hodgkin Study Group. Leukemia. 2020 Mar;34(3):953-956. doi: 10.1038/s41375-019-0609-3. Epub 2019 Oct 21. No abstract available. PMID 31636342
- [Derived] Eichenauer DA, Fuchs M, Pluetschow A, Klimm B, Halbsguth T, Boll B, von Tresckow B, Nogova L, Borchmann P, Engert A. Phase 2 study of rituximab in newly diagnosed stage IA nodular lymphocyte-predominant Hodgkin lymphoma: a report from the German Hodgkin Study Group. Blood. 2011 Oct 20;118(16):4363-5. doi: 10.1182/blood-2011-06-361055. Epub 2011 Aug 9. PMID 21828141